CLINICAL TRIAL: NCT03925389
Title: Functional and Aesthetic Outcome Analysis in External Septorhinoplasty
Brief Title: Outcome Analysis in Septorhinoplasty
Status: Recruiting | Type: Observational
Sponsor: FRANK DECLAU (Other)
Collaborators: Universiteit Antwerpen (Other); Gasthuis Zusters Antwerpen (Other)
Responsible Party: Sponsor-Investigator, FRANK DECLAU, Head of Otolaryngology Department, Visiting professor, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Other Study IDs: FDSV02
Record Dates: First submitted 2019-04-13; First posted 2019-04-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Rhinoplasty; Nasal Obstruction; Esthetics
Keywords: Nasal function; Septorhinoplasty; Patient-reported outcome; Rhinomanometry; Acoustic Rhinometry; Peak Nasal Inspiratory Flow; Esthetics
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: External septorhinoplasty — A surgical procedure to repair defects or deformities of both the nasal septum and the external nasal pyramid through an external incision at the columella.

SUMMARY:
A prospective observational cohort study that measures pre- and postoperative outcome of septorhinoplasty by means of patient-related outcome measures (PROMS: NOSE, FACE-Q, Utrecht Questionnaire, SCHNOS and BDDQ-AS) as well as with functional tests (NAR, AR, PNIF).

DETAILED DESCRIPTION:
Introduction:

In an ENT setting, septorhinoplasty is frequently performed for both functional and aesthetic reasons. Therefore, pre- and postoperative evaluation of patients' 'total' satisfaction regarding their nasal appearance and functional result is paramount.

Objectives:

To measure the pre- and postoperative functional and aesthetic outcome in patients undergoing an external septorhinoplasty.

Design, setting, participants:

A prospective observational, longitudinal outcome cohort study in a single private hospital centre is set up. All participants are patients undergoing an external septorhinoplasty for functional and aesthetic reasons.

Exposures:

The Nasal Obstruction Symptom Evaluation scale (NOSE), Utrecht questionnaire, the FACE-Q Satisfaction With Nose, FACE-Q Satisfaction With Nostrils, SCHNOS score and BDDQ-AS score, are administered to patients preoperatively and at 3, 6 and 12 months postoperatively. Also functional tests (nasal anterior rhinomanometry (NAR), Peak nasal inspiratory flow (PNIF) and acoustic rhinometry (AR) will be performed preoperatively and postoperatively at 6 and 12 months. Patient demographics, nasal history, and outcomes will be analyzed.

Main outcome and measures:

The primary outcome will measure longitudinal postoperative changes in nasal obstruction and aesthetic satisfaction:

* Change between pre- and postoperative results of NOSE and FACE-Q questionnaires, Utrecht questionnaire, SCHNOS and BDDQ-AS score (time frame: at inclusion and at 3, 6 and 12 months postoperatively)
* Change between pre- and postoperative values of NAR, PNIF and acoustic rhinometry (time frame: at inclusion and at 6 and 12 months postoperatively)

Secondary outcome

* Correlation between PROMS and functional tests
* Correlation between change in functional tests and the surgical methods used

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* Patients eligible for external septorhinoplasty: patients seen in consultation because of nasal obstruction were evaluated. Patients who had symptoms of nasal obstruction for at least 1 year that were the result of an identifiable anatomical cause such as septal deviation, turbinate hypertrophy, internal valve collapse, or external valve collapse were included in the study.

Exclusion Criteria:

* < 18 years
* mental or physical incapacity to answer the questionnaires
* nasal fracture or surgery in the past year
* nasal cocaine use in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants eligible for external septorhinoplasty will consecutively be enrolled in the study according to CONSORT guidelines
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of pre- and postoperative changes in aesthetic satisfaction using FACE-Q (TM) questionnaire | 12 months
  Change between pre- and postoperative results of FACE-Q questionnaire.
  • FACE-Q (TM): Two items of the FACE-Q (TM) instrument (satisfaction with nose and satisfaction with nostrils) are used:
  * Subscale 'Satisfaction of the nostrils': score from 0 (very unsatisfied) to 100 (very satisfied).
  * Subscale 'Satisfaction of the nose': score from 0 (very unsatisfied) to 100 (very satisfied).
Measurement of pre- and postoperative changes in nasal obstruction using NOSE questionnaire | 12 months
  Change between pre- and postoperative results of NOSE questionnaire.
  • NOSE (Nasal Obstruction and Septoplasty Effectiveness Scale): scale from 0 (no nasal obstruction) to 100 (severe nasal obstruction).
Measurement of pre- and postoperative changes in nasal obstruction using acoustic rhinometry | 12 months
  Change between pre- and postoperative acoustic rhinometry:
  •AR (acoustic rhinometry): minimal cross-sectional area (cm2) (MCA) is measured for each nostril separately.
Measurement of pre- and postoperative changes in nasal obstruction using peak nasal inspiratory flow: | 12 months
  Change between pre- and postoperative peak nasal inspiratory flow:
  •PNIF (peak nasal inspiratory flow): peak nasal inspiratory flow (l/min) is measured for each nostril separately.
Measurement of pre- and postoperative changes in nasal obstruction using rhinomanometry | 12 months
  Change between pre- and postoperative rhinomanometry :
  •NAR(nasal anterior rhinomanometry) : nasal airflow at 150 Pa is recorded for each nostril separately (ml/sec).
Measurement of pre- and postoperative changes in aesthetic satisfaction Utrecht Questionnaire: 6 items scale: - 5 items with Likert scale from 5 (not at all) to 25 very (often) - 1 item: VAS score from 0 (very ugly) to 10 (very nice) | 12 months
  Change between pre- and postoperative results of Utrecht questionnaire.
Measurement of pre- and postoperative changes in aesthetic satisfaction and nasal obstruction using the SCHNOS Questionnaire | 12 months
  Change between pre- and postoperative results of SCHNOS questionnaire. 10 items scale from 0 (no problem) to 5 (severe problem).
Measurement of pre- and postoperative changes in aesthetic satisfaction using the BDD (Body Dysmorphic Disorder) Questionnaire. 7 items scale: item 1-2 : dichotomous (yes/no) Item 3-6: 1(mild) to 5 (extreme) Item 7: dichotomous (yes/no) | 12 months
  Change between pre- and postoperative results of BDD questionnaire.

SECONDARY OUTCOMES:
Correlation between NOSE questionnaire and nasal functional tests | 12 months
  Correlation between:
  NOSE (Nasal Obstruction and Septoplasty Effectiveness Scale): scale from 0 (no nasal obstruction) to 100 (severe nasal obstruction).
  and: NAR(nasal active rhinomanometry) : nasal airflow at 150 Pa is recorded for each nostril separately (ml/sec).
  PNIF (peak nasal inspiratory flow): peak nasal inspiratory flow (l/min) is measured for each nostril separately.
  AR (acoustic rhinometry): minimal cross-sectional area (cm2) (MCA) is measured for each nostril.
Correlation between change of nasal functional tests and surgical methods | 12 months
  NAR(nasal active rhinomanometry) : nasal airflow at 150 Pa is recorded for each nostril separately (ml/sec).
  PNIF (peak nasal inspiratory flow): peak nasal inspiratory flow (l/min) is measured for each nostril separately.
  AR (acoustic rhinometry): minimal cross-sectional area (cm2) (MCA) is measured for each nostril.
  and: surgical data acquired from the operative report from each patient: technical procedures undertaken to improve nasal obstruction by addressing the anatomic structures that comprise the internal and/or external nasal valves.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Declau, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Dept. Otorhinolaryngology, H&N Surgery, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pingnet L, Verkest V, Fransen E, Declau F. Dutch Translation and Validation of the FACE-Q Rhinoplasty Module. Facial Plast Surg. 2021 Jun;37(3):296-301. doi: 10.1055/s-0040-1721099. Epub 2021 Jan 27. PMID 33506453
- [Background] Valérie Verkest, Laura Pİngnet, Erik Fransen, Frank Declau. Analysis of functional and aesthetic outcomes in external septorhinoplasty: study protocol. B-ENT 2020; 16: 45-50 DOI: 10.5152/B-ENT.2020.19125
- [Background] Declau F, Pingnet L, Verkest V, Hansen T. Cross-Cultural Evaluation of the Dutch FACE-Q Rhinoplasty Questionnaires Using Rasch Analysis. Aesthet Surg J. 2021 Nov 12;41(12):NP1916-NP1930. doi: 10.1093/asj/sjab217. PMID 33945612
- [Background] Verkest V, Pingnet L, Fransen E, Declau F. Multidimensionality of Patient-Reported Outcome Measures in Rhinoplasty Satisfaction. Facial Plast Surg. 2022 Oct;38(5):468-476. doi: 10.1055/a-1760-1422. Epub 2022 Feb 3. PMID 35114725
- [Background] Verkest V, Pingnet L, Fransen E, Declau F. Piezo-assisted Turbinoplasty Versus Partial Turbinectomy in External Septorhinoplasty: A Prospective Comparative Study in 100 Patients. Aesthetic Plast Surg. 2022 Jun;46(3):1323-1331. doi: 10.1007/s00266-021-02662-0. Epub 2022 Jan 13. PMID 35022839
- [Background] Pingnet L, Verkest V , Saltychev M , Most SP , Declau F. Translation and Validation of the Standardized Cosmesis and Health Nasal Outcomes Survey in Dutch. B-ENT 2022; 18: 170-175. doi: 10.5152/B-ENT.2022.22910.